CLINICAL TRIAL: NCT00685100
Title: Retinal Effects After Combined Photodynamic Therapy (PDT) With Intravitreal Triamcinolone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Priv.Doz. Dr. Stefan Sacu, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2008-05

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: IVTA; CNV; age-related macular degeneration; PDT
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — 1-phenyl-3,3-dimethyltriazene

INTERVENTIONS:
Other: PDT plus intravitreal triamcinolone — PDT plus intravitreal triamcinolone

SUMMARY:
Background: To identify characteristic morphological changes of the retina, their change over time and the association with visual function after combined photodynamic therapy (PDT) and intravitreal triamcinolone (IVTA).

Methods: In this retrospective study, 40 patients (40 eyes) were treated with PDT and same day IVTA. Optical coherence tomography (OCT), fluorescein angiography (FA) and evaluation of distance visual acuity (VA) were performed. Main outcome measures were the anatomical changes within intra- and subretinal compartments and their detailed analysis and grading.

ELIGIBILITY:
Inclusion Criteria:

* cnv secondary to age related macular degeneration

Exclusion Criteria:

* glaucoma, diabetic retinopathy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
visual acuity, central retinal thickness (CRT), choroidal perfusion and macular sensitivity (MS) | Day 1, Week 1, 4 and 12
  "Changes in macular sensitivity after reduced fluence photodynamic therapy combined with intravitreal triamcinolone" Mean DLT decreased from 4.71 dB at baseline to 3.45 dB after 12 months in the SPDT + IVTA group (mean decrease 1.26 dB; p > 0.05) and from 5.42 dB to 4.92 dB in the RPDT + IVTA group (mean decrease 0.5 dB; p > 0.05). Absolute and relative scotoma sizes remained stable in both groups at 12 months (mean change 0 and -0.6 test-points; p > 0.05). Mean DLT values and absolute scotoma sizes correlated well with early and late leakage areas in FA (r = -0.45 to -0.80, p < 0.02).
  With regard to MS, RPDT + IVTA did not show significant benefits over SPDT + IVTA at 12 months. Macular sensitivity correlated well with angiographic outcomes.
visual acuity, central retinal thickness (CRT), choroidal perfusion and macular sensitivity (MS) | Day 1, week 1, 4 and 12
  "Reduced fluence versus standard photodynamic therapy in combination with intravitreal triamcinolone: short-term results of a randomised study" Baseline characteristics were well balanced in both groups (p>0.05). At week 12, patients in group A had a mean loss of -3.7 letters compared with a gain of 3.4 letters in group B (p = 0.04, between both groups). Both treatment groups showed a similar course regarding CRT as well as MS (p>0.05). In 70% (14/20) of group A and 15% (3/20) of group B, a choroidal hypoperfusion in the area of treatment was observed after treatment (p<0.001). In 70% of group A and 55% of group B, a repeat treatment was indicated at week 12 (p = 0.55).
  At month 3, the rPDT+IVTA group showed a significantly better visual outcome, less alteration of the choroid and a trend for lower recurrence rate than the sPDT+IVTA group. Further follow-up of this study will provide information on long-term functional results and treatment durability.